CLINICAL TRIAL: NCT02460315
Title: Early Versus Late Cholecystectomy After Clearance of Common Bile Duct Stones by Endoscopic Retrograde Cholangiopancreatography
Brief Title: Early Versus Late Cholecystectomy After Clearance of Common Bile Duct Stones
Acronym: ERCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ayman El Nakeeb, Gastroenterology surgical center, mansoura university, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: timing of cholecystectomy
Record Dates: First submitted 2015-05-22; First posted 2015-06-02 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2013-05

CONDITIONS: Gallbladder and Bile Duct Calculi
Keywords: time of cholecystectomy after ERCP

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- early cholecystectomy (Active Comparator): group (A) will be managed by early laparoscopic cholecystectomy after clearness ERCP
  Interventions: Procedure: early cholecystectomy
- late cholecystectomy (Active Comparator): group (B) will be managed by late LC one month after ERCP.
  Interventions: Procedure: late cholecystectomy

INTERVENTIONS:
Procedure: early cholecystectomy — Those patients are primarily managed by endoscopic sphincterotomy and stone extraction for management of CBD stones. Then, the study population will be divided into 2 groups; group 1 will be managed by early laparoscopic cholecystectomy (LC) within 3 days after ERCP
  Other Names: G 1
  Arms: early cholecystectomy
Procedure: late cholecystectomy — Those patients are primarily managed by endoscopic sphincterotomy and stone extraction for management of CBD stones. Then, the study population will be divided into 2 groups; group 2 will be managed by late LC one month after ERCP.
  Other Names: G 2
  Arms: late cholecystectomy

SUMMARY:
Approximately 10-15% of all patients with gallstones have coexisting common bile duct (CBD) stones. However CBD stones can also be formed in the absence of gallbladder stones. The current standard of treatment for calcular obstructive jaundice is endoscopic removal of the stones. Endoscopic sphincterotomy (ES) is widely accepted as the treatment of choice for patients with CBDS. Stone extraction is successful in up to 97% of patients The time interval between ERCP and laparoscopic cholecystectomy (LC) is a matter of debate that may vary from days to months. Some retrospective and other prospective studies have investigated this issue without sharp clue or definite conclusion This study planned to compare early LC (within admission) versus late LC (after 1 month) after ERCP as regard technical difficulties and surgical outcomes.

DETAILED DESCRIPTION:
The aim is comparing early versus delayed laparoscopic cholecystectomy after endoscopic retrograde cholangiopancreatography in patients with gall bladder stones and calcular obstructive jaundice as regards operative difficulties, conversion rate, signs of inflammation, degree of adhesions, blood loss, postoperative morbidity, and hospital stay. Moreover, bacterial examination of bile and culture sensitivity test for assessment of bacterial colonization and relate the degree of colonization to timing of laparoscopic cholecystectomy after endoscopic retrograde cholangiopancreatography, to decide upon the optimal timing for the surgery.

The study population will be divided into 2 groups; group (A) will be managed by early laparoscopic cholecystectomy (LC) within 3 days after ERCP and group (B) will be managed by late LC one month after ERCP.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CBD stone and treated by ERCP

Exclusion Criteria:

* Patient unfit for surgery,
* Pregnant patients,
* Patients with severe malnutrition,
* Patients with liver cirrhosis,
* Patients in whom endoscopic management of CBD stones failed
* Patients who experienced pancreatitis or perforation as a complication of the endoscopic management of CBD stones
* Patients who underwent previous upper abdominal surgeries
* Mentally retarded patients.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-05; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
conversion rate to open | 1 day
  number of patients underwent conversion to open

SECONDARY OUTCOMES:
signs of inflammation (redness, pus) | 30 days
  signs of inflammation redness, pus, wall thickness
postoperative morbidity | 1 days
  postoperative morbidity
degree of adhesion (mild,moderate, severe) | 1 days
  degree of adhesions

CONTACTS AND LOCATIONS:
Overall Officials: Ayman El Nakeeb, MD, Principal Investigator — Mansoura University

REFERENCES:
- [Result] Bostanci EB, Ercan M, Ozer I, Teke Z, Parlak E, Akoglu M. Timing of elective laparoscopic cholecystectomy after endoscopic retrograde cholangiopancreaticography with sphincterotomy: a prospective observational study of 308 patients. Langenbecks Arch Surg. 2010 Aug;395(6):661-6. doi: 10.1007/s00423-010-0653-y. Epub 2010 Jun 6. PMID 20526779
- [Result] Mo LR, Chang KK, Wang CH, Yau MP, Yang TM. Preoperative endoscopic sphincterotomy in the treatment of patients with cholecystocholedocholithiasis. J Hepatobiliary Pancreat Surg. 2002;9(2):191-5. doi: 10.1007/s005340200017. PMID 12140605
- [Result] Schiphorst AH, Besselink MG, Boerma D, Timmer R, Wiezer MJ, van Erpecum KJ, Broeders IA, van Ramshorst B. Timing of cholecystectomy after endoscopic sphincterotomy for common bile duct stones. Surg Endosc. 2008 Sep;22(9):2046-50. doi: 10.1007/s00464-008-9764-8. Epub 2008 Feb 13. PMID 18270768